CLINICAL TRIAL: NCT00605228
Title: A Randomised, Multicentre, Single-Blind, Phase IV Study, of the Efficacy, Safety, and Acceptability of Moviprep® Versus Colopeg® in Colonoscopy Preparation.
Brief Title: A Phase IV Study, of the Efficacy, Safety, and Acceptability of Moviprep® Versus Colopeg® in Colonoscopy Preparation
Acronym: NORMO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Norgine (Industry)
Collaborators: International Clinical Trials Association (Other)
Responsible Party: Cécile DUGUE Medical Director, Norgine Pharma
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRL994-02/2006 (FFS)
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2008-01

CONDITIONS: Gastrointestinal Diseases
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — MoviPrep

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: MOVIPREP
- 2 (Active Comparator)
  Interventions: Drug: COLOPEG

INTERVENTIONS:
Drug: MOVIPREP — 2L Drug
  Arms: 1
Drug: COLOPEG — 4L Drug
  Arms: 2

SUMMARY:
Primary:

- To demonstrate the superiority of Moviprep® versus Colopeg® in gut cleansing prior to colonoscopy.

Secondary:

* To assess the safety of Moviprep® versus Colopeg®.
* To assess acceptability of Moviprep® versus Colopeg®.

DETAILED DESCRIPTION:
Primary efficacy analysis will be performed on the ITT population. Secondary efficacy analysis will be performed on both ITT and PP sets. Results will be summarised by treatment and age (overall, 18-35, 36-49, 50-74 and 75-85 years old) and provided in individual data listings.

Safety analysis will be performed on the safety set (ITT population). Safety data of all patients exposed will be summarised by treatment and age (overall, 18-35, 36-49, 50-74 and 75-85 years old).

Acceptability analysis will be performed on the ITT population. Acceptability data of all patients will be summarised by treatment and age (overall, 18-35, 36-49, 50-74 and 75-85 years old).

ELIGIBILITY:
Inclusion Criteria:

1. The patient's written informed consent must be obtained prior to inclusion.
2. Male or female, outpatients between 18 and 85 years old with an indication to colonoscopy.
3. Willing and able to complete the entire procedure and to comply with study instructions.
4. Females of childbearing potential must employ an adequate method of birth control.

Exclusion Criteria:

1. Age < 18 or > 85 years old,
2. Ileus,
3. Suspected intestinal occlusion or perforation,
4. Toxic megacolon with severe inflammation conditions of intestinal tract (patients with Crohn's Disease or Ulcerative Colitis included),
5. Gastroparesis,
6. Congestive heart failure NYHA III or IV,
7. Documented Carcinoma or any other colic disease leading to a fragile mucosa,
8. Documented severe renal insufficiency history
9. Known hypersensitivity to MoviPrep®, Colopeg® or to any of their components (PEG, ascorbic acid etc.),
10. Known deficiency in G6PD and/or phenylketonuria,
11. Concurrent participation in an investigational drug/device study or participation within 30 days of study entry,
12. Females who are pregnant, or planning a pregnancy. Females of child bearing potential not using reliable methods of birth control,
13. Clinically significant laboratory abnormality or disease which, in the opinion of the investigator, will create a risk for the patient, obscure the effects of study treatment or interfere with study results.
14. Vulnerable patients (protected by the law) and those admitted to a sanitary/social institution according to Art.L-1121-6 of the French Public Health Code.

    -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2007-05; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
the proportion of patients with successful colon cleansing as judged by blinded reviewers on the basis of videotapes recorded during the colonoscopy [the blinded reviewers will grade the colon cleansing only once] | 1 day

SECONDARY OUTCOMES:
the proportion of patients with successful colon cleansing as judged by the colonoscopist, the colonic segment cleansing score as assessed by the colonoscopist and the blinded reviewers and Aronchick global score as assessed by blinded reviewers. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Thierry PONCHON, MD, Principal Investigator — HOPITAL EDOUARD HERRIOT
Locations (21):
- France (21):
  - Centre Hospitalier Du Mans, Le Mans, Lemans
  - Service d'Hépato-Gastroentérologie, CHRU NANCY, HOPITAL DE BRABOIS, Nancy, Nancy
  - Service de Gastroentérologie du Pr. LEREBOURS, HOPITAL CHARLES NICOLLE, Rouen, Rouen
  - Cabinet de gatsro-entérologie, Anglet
  - Cabinet de gastroentérologie, Aubagne
  - Service de Gastroentérologie,CENTRE HOSPITALIER d'AVIGNON, Avignon
  - Clinique de La Châtaigneraie, Beaumont
  - Cabinet de gastro-entérologie, Bordeaux
  - Clinique Saint Martin, Caen
  - Service de Gastroentérologie du Dr. Chousterman, HOPITAL INTERCOMMUNAL, Créteil
  - Centre Des Maladies Du Foie Et de L'Appareil Digestif, Irigny
  - Cabinet de gastroentérologie, Les Sables-d'Olonne
  - Cabinet Medical Jemmapes, Lille
  - Service de Gastroentérologie, HOPITAL DE L'ARCHET, Nice
  - Service de Gastro-Entérologie, HÔPITAL GEORGES POMPIDOU, Paris
  - Service de Gastroentérologie du Pr. MARTEAU, HÔPITAL LARIBOISIERE, Paris
  - Hopital F. Mitterand, Pau
  - Polyclinique Courlancy, Reims
  - Service des Maladies de l'Appareil Digestif, Centre Hospitalier Régional et Universitaire, Rennes
  - Clinique Saint Jean Languedoc, Toulouse
  - Service de Gastro-Entérologie, HOPITAL TROUSSEAU CHRU de Tours, Tours

REFERENCES:
- [Background] Bitoun A, Ponchon T, Barthet M, Coffin B, Dugue C, Halphen M; Norcol Group. Results of a prospective randomised multicentre controlled trial comparing a new 2-L ascorbic acid plus polyethylene glycol and electrolyte solution vs. sodium phosphate solution in patients undergoing elective colonoscopy. Aliment Pharmacol Ther. 2006 Dec;24(11-12):1631-42. doi: 10.1111/j.1365-2036.2006.03167.x. Epub 2006 Nov 10. PMID 17094774